CLINICAL TRIAL: NCT03327090
Title: The Effect of the Kinesio Tape on the Muscle Power Performance of Elite Weightlifters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB- PGS- 2015- 03- 205
Record Dates: First submitted 2017-09-23; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Muscle Power Performance
Keywords: Olympic Weightlifting; Taping; Muscles Facilitation; Jumps

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Kinesio Tape (Experimental): The Kinesio Tape original brand was used in this study (Kinesio® Tex GoldTM finger print, black, Georgia, Albuquerque). The application of the experimental Kinesio Tape was as Dr. Kenzo Kase demonstration for muscle facilitation (Kase. et al., 2003):
  1. Gluteal maximus muscle.
  2. Quadriceps muscle.
  3. Gastrocnemius muscle and soleus muscle (triceps surae).
  The tape was in tension (15%- 35%) and the muscles were stretched during the application.
  Interventions: Other: Kinesio Tape original brand (Kinesio® Tex GoldTM finger print, black, Georgia, Albuquerque).
- Sham Kinesio Tape (Sham Comparator): Same tape brand was used, but different application techniques were utilized for the three muscles.
  1. Gluteal maximus muscle.
  2. Quadriceps muscle.
  3. Gastrocnemius muscle and soleus muscle (triceps surae).
  There were no tension on the tape and no muscle stretching during the application.
  Interventions: Other: Kinesio Tape original brand (Kinesio® Tex GoldTM finger print, black, Georgia, Albuquerque).

INTERVENTIONS:
Other: Kinesio Tape original brand (Kinesio® Tex GoldTM finger print, black, Georgia, Albuquerque). — Kinesio Tape: An elastic therapeutic tape, which mimics the skin's thickness. It is a cotton, porous fabric and acrylic adhesive, which is non-medicated and free of latex. The Kinesio Tape is applied in a specific manner to enhance muscle function, increase circulation, decrease pain and improve proprioception.

SUMMARY:
This study is aimed to investigate the effect of the Kinesio Tape facilitation technique on the muscle power performance of elite weightlifters.

DETAILED DESCRIPTION:
Most sportsmen require the power of muscles for their performance. Weightlifting exercises such as the snatch or clean and jerk and their variations are frequently included in the power training programs of athletes who contest or participate in sports that need muscle power. The weightlifting exercises require athletes to accelerate the weight throughout the whole second pull phase, causing the barbell to be raised overhead and the athlete's body into the air, a movement in which the feet leave the platform. Furthermore, the movement patterns of the weightlifting exercises are mostly considered to be similar to athletic movements in different sports such as jumping and sprinting in soccer and basketball. Empirically, the kinetic qualities of the second pull phase are similar in both weightlifting and jumping movements. The role of the sport physical therapist is not restricted only to rehabilitation and injuries prevention, but they can also contribute to the performance of the athletes in a different aspect. Therefore, finding tools which may improve the muscle power of the weightlifters could increase the success in performing the sport-specific movements with higher loads. This could make the difference between winning or losing a competition. Thus, if it could be proven that the Kinesio Tape has the capability to improve muscle power, it could be used as a tool by the physiotherapist, either for enhancing the athlete's performance or for accelerating the last stage of the rehabilitation and, therefore, decreasing the number of absent days of athletes from training or matches due to injury.

ELIGIBILITY:
Inclusion Criteria:

* 46 Male weightlifters from 18-35 years old.
* Weightlifters who playing at national weightlifting level.

Exclusion Criteria:

* Musculoskeletal injuries or surgery that may affect performance in the last 6 weeks prior to the study as reported by participant.
* Any neurological problem that may affect performance as reported by the participant.
* Known adverse reactions to taping.
* Any systemic diseases that affect the performance as reported by participant.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2016-03-13 (Actual); Study Completion 2016-03-13 (Actual)

PRIMARY OUTCOMES:
Single leg vertical countermovement jump. | Data was collected on January 7, 2016 up to March 13, 2016 (an average of three months) in which the collection of the data was finished.
  Participants were performed three vertical jump attempts with a counter-movement.
Single leg horizontal countermovement jump | Data was collected on January 7, 2016 up to March 13, 2016 (an average of three months) in which the collection of the data was finished.
  Participants were performed three horizontal jump attempts with a counter-movement.

SECONDARY OUTCOMES:
Estimated peak power. | The estimated peak power was calculated and reviewed at the end of data collection on March 13, 2016 up to April 7, 2016 ( an average of one month).
  A predictive equation to calculate an anaerobic power output from the vertical jump displacement.

CONTACTS AND LOCATIONS:
Overall Officials: Majed A Al-Abbad, MSc, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- University of Dammam, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No